CLINICAL TRIAL: NCT04853017
Title: First in Human Phase 1 Trial of ELI-002 Immunotherapy as Treatment for Subjects With Kirsten Rat Sarcoma (KRAS) Mutated Pancreatic Ductal Adenocarcinoma and Other Solid Tumors
Brief Title: A Study of ELI-002 in Subjects With KRAS Mutated Pancreatic Ductal Adenocarcinoma (PDAC) and Other Solid Tumors
Acronym: AMPLIFY-201
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Elicio Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ELI-002-001
Record Dates: First submitted 2021-04-16; First posted 2021-04-21 (Actual); Results first posted 2025-01-17 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Minimal Residual Disease; KRAS G12D; KRAS G12R; NRAS G12D; NRAS G12R; Pancreatic Ductal Adenocarcinoma; Colorectal Cancer; Non-small Cell Lung Cancer; Ovarian Cancer; Cholangiocarcinoma; Bile Duct Cancer; Gallbladder Carcinoma
Keywords: Minimal residual disease (MRD); Kirsten rat sarcoma (KRAS); Neuroblastoma ras viral oncogene homolog (NRAS); Pancreatic ductal adenocarcinoma (PDAC); Colorectal cancer (CRC); Colon cancer; Rectal cancer; Non-small-cell lung cancer (NSCLC); Mucinous Ovarian cancer; Cholangiocarcinoma (CCA); Bile duct cancer; Gallbladder carcinoma; Immunotherapy; Vaccine therapy; Adjuvant therapy; circulating tumor DNA (ctDNA)
MeSH Terms: conditions — Neoplasm, Residual; Colorectal Neoplasms; Carcinoma, Non-Small-Cell Lung; Ovarian Neoplasms; Cholangiocarcinoma; Bile Duct Neoplasms; Gallbladder Neoplasms; Colonic Neoplasms; Rectal Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- ELI-002 2P Cohort 1 (Experimental): ELI-002 2P Amph-CpG-7909 (0.1 mg) admixed with Amph modified KRAS peptides (Amph-G12D and Amph-G12R) administered via subcutaneous (SC) injection weekly for 4 consecutive weeks, followed by bi-weekly injections over 4 weeks, during the Immunization period; additional SC injections weekly for 4 consecutive weeks during the Booster Period (the two periods are separated by 3 months of no dosing)
  Interventions: Drug: ELI-002 2P
- ELI-002 2P Cohort 2 (Experimental): ELI-002 2P Amph-CpG-7909 (0.5 mg) admixed with Amph modified KRAS peptides (Amph-G12D and Amph-G12R) administered via SC injection weekly for 4 consecutive weeks, followed by bi-weekly injections over 4 weeks, during the Immunization period; additional SC injections weekly for 4 consecutive weeks during the Booster Period (the two periods are separated by 3 months of no dosing)
  Interventions: Drug: ELI-002 2P
- ELI-002 2P Cohort 3 (Experimental): ELI-002 2P Amph-CpG-7909 (2.5 mg) admixed with Amph modified KRAS peptides (Amph-G12D and Amph-G12R) administered via SC injection weekly for 4 consecutive weeks, followed by bi-weekly injections over 4 weeks, during the Immunization period; additional SC injections weekly for 4 consecutive weeks during the Booster Period (the two periods are separated by 3 months of no dosing)
  Interventions: Drug: ELI-002 2P
- ELI-002 2P Cohort 4 (Experimental): ELI-002 2P Amph-CpG-7909 (5.0 mg) admixed with Amph modified KRAS peptides (Amph-G12D and Amph-G12R) administered via SC injection weekly for 4 consecutive weeks, followed by bi-weekly injections over 4 weeks, during the Immunization period; additional SC injections weekly for 4 consecutive weeks during the Booster Period (the two periods are separated by 3 months of no dosing)
  Interventions: Drug: ELI-002 2P
- ELI-002 2P Cohort 5 (Experimental): ELI-002 2P Amph-CpG-7909 (10.0 mg) admixed with Amph modified KRAS peptides (Amph-G12D and Amph-G12R) administered via SC injection weekly for 4 consecutive weeks, followed by bi-weekly injections over 4 weeks, during the Immunization period; additional SC injections weekly for 4 consecutive weeks during the Booster Period (the two periods are separated by 3 months of no dosing)
  Interventions: Drug: ELI-002 2P

INTERVENTIONS:
Drug: ELI-002 2P — Amph-CpG-7909 admixed with Amph modified KRAS peptides (Amph-G12D and Amph-G12R) administered via SC injection weekly for 4 consecutive weeks, followed by bi-weekly injections over 4 weeks, during the Immunization Period; additional SC injections weekly for 4 consecutive weeks during the Booster Period (the two periods are separated by 3 months of no dosing)

SUMMARY:
This is a Phase 1 study to assess the safety and efficacy of ELI-002 immunotherapy (a lipid-conjugated immune-stimulatory oligonucleotide [Amph-CpG-7909] plus a mixture of lipid-conjugated peptide-based antigens [Amph-Peptides]) as adjuvant treatment of minimal residual disease (MRD) in subjects with KRAS/neuroblastoma ras viral oncogene homolog (NRAS) mutated PDAC or other solid tumors.

DETAILED DESCRIPTION:
This is a Phase 1 dose escalation study in which ELI-002 2P (Amph modified KRAS peptides, Amph-G12D and Amph-G12R admixed with admixed Amph-CpG-7909) will be evaluated, with plans to transition to the ELI-002 7P drug product containing all 7 Amph-Peptides (G12D, G12R, G12V, G12A, G12C, G12S, G13D) in future clinical trials.

The study is an open-label, dose-escalation, 3+3 design in which approximately 18 subjects will be treated in 3 planned dose level cohorts. Increasing doses of Amph-CpG-7909 will be evaluated sequentially. Additional cohorts may be added to explore intermediate or higher dose levels based on cumulative safety review and preliminary review of pharmacodynamic responses. Safety and pharmacodynamic data will be evaluated and a recommended Phase 2 dose (RP2D) will be determined in consideration of a maximum tolerated dose (MTD) if observed.

ELIGIBILITY:
Inclusion Criteria:

* KRAS/NRAS mutated (G12D or G12R) solid tumor
* Positive for circulating tumor DNA (ctDNA) and/or elevated serum tumor biomarker despite prior standard therapy including surgery and chemotherapy/radiation therapy where applicable
* Screening CT is negative for recurrent disease
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1

Exclusion Criteria:

* Presence of tumor mutations where specific therapy is approved, and the patient is able to receive the approved therapy
* Known brain metastases
* Use of immunosuppressive drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2021-10-04 (Actual); Primary Completion 2023-01-26 (Actual); Study Completion 2024-09-24 (Actual)

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - City of Hope, Duarte, California
  - University of California Los Angeles, Los Angeles, California
  - University of Colorado, Aurora, Colorado
  - University of Iowa, Iowa City, Iowa
  - Massachusetts General Hospital, Boston, Massachusetts
  - Washington University School of Medicine, St Louis, Missouri
  - Northwell Health, Lake Success, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Tennessee Oncology - Centennial Clinic, Nashville, Tennessee
  - The University of Texas MD Anderson Cancer Center, Houston, Texas

REFERENCES:
- [Derived] Wainberg ZA, Weekes CD, Furqan M, Kasi PM, Devoe CE, Leal AD, Chung V, Perry JR, Kheoh T, McNeil LK, Welkowsky E, DeMuth PC, Haqq CM, Pant S, O'Reilly EM. Lymph node-targeted, mKRAS-specific amphiphile vaccine in pancreatic and colorectal cancer: phase 1 AMPLIFY-201 trial final results. Nat Med. 2025 Nov;31(11):3648-3653. doi: 10.1038/s41591-025-03876-4. Epub 2025 Aug 11. PMID 40790272
- [Derived] Pant S, Wainberg ZA, Weekes CD, Furqan M, Kasi PM, Devoe CE, Leal AD, Chung V, Basturk O, VanWyk H, Tavares AM, Seenappa LM, Perry JR, Kheoh T, McNeil LK, Welkowsky E, DeMuth PC, Haqq CM, O'Reilly EM. Lymph-node-targeted, mKRAS-specific amphiphile vaccine in pancreatic and colorectal cancer: the phase 1 AMPLIFY-201 trial. Nat Med. 2024 Feb;30(2):531-542. doi: 10.1038/s41591-023-02760-3. Epub 2024 Jan 9. PMID 38195752

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | ELI-002 2P Cohort 1 | ELI-002 2P Cohort 2 | ELI-002 2P Cohort 3 | ELI-002 2P Cohort 4 | ELI-002 2P Cohort 5
Started | 3 | 6 | 5 | 5 | 6
Completed | 1 | 2 | 2 | 3 | 3
Not Completed | 2 | 4 | 3 | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- ELI-002 2P Cohort 1: ELI-002 2P Amph-CpG-7909 (0.1 mg) admixed with Amph modified KRAS peptides (Amph-G12D and Amph-G12R) administered via SC injection weekly for 4 consecutive weeks, followed by bi-weekly injections over 4 weeks, during the Immunization period; additional SC injections weekly for 4 consecutive weeks during the Booster Period (the two periods are separated by 3 months of no dosing)
  ELI-002 2P: Amph-CpG-7909 admixed with Amph modified KRAS peptides (Amph-G12D and Amph-G12R) administered via SC injection weekly for 4 consecutive weeks, followed by bi-weekly injections over 4 weeks, during the Immunization Period; additional SC injections weekly for 4 consecutive weeks during the Booster Period (the two periods are separated by 3 months of no dosing)
- Total: Total of all reporting groups
Arm/Group | ELI-002 2P Cohort 1 | ELI-002 2P Cohort 2 | ELI-002 2P Cohort 3 | ELI-002 2P Cohort 4 | ELI-002 2P Cohort 5 | Total
Number analyzed (Participants) | 3 | 6 | 5 | 5 | 6 | 25
Age, Continuous [Median (Full Range); unit: years] | 50.0 [47 to 61] | 54.5 [37 to 69] | 67.0 [63 to 77] | 67.0 [47 to 75] | 59.0 [48 to 69] | 61.0 [37 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 5 | 4 | 3 | 1 | 15
  Male | 1 | 1 | 1 | 2 | 5 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 0 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0
  White | 2 | 5 | 4 | 5 | 5 | 21
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1 | 0 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 3 | 6 | 5 | 5 | 6 | 25
Pancreatic ductal adenocarcinoma diagnosis [Count of Participants; unit: Participants] | 1 | 4 | 5 | 4 | 6 | 20
Disease stage at screening [Count of Participants; unit: Participants] — Cancer staging per the American Joint Committee on Cancer is determined based on tumor size, spread to lymph nodes, and spread to other parts of the body (metastases). Stage 1: a small tumor that is contained in one area and has not spread. Stage 2: a larger tumor that has possibly spread to nearby lymph nodes. Stage 3: a tumor that has spread to lymph nodes or nearby tissue. Stage 4: a tumor that has spread to distant sites in the body (in this trial, Stage 4 disease was oligometastatic with < 3 lesions in one organ). Generally, progressively higher stages have progressively worse outcomes.
  Participants
    Stage I, II | 1 | 2 | 3 | 1 | 1 | 8
    Stage III, IV | 2 | 4 | 2 | 4 | 5 | 17

OUTCOME MEASURES:

1. Primary Outcome: The Participant Incidence of Treatment-emergent Adverse Events Considered by the Investigator as Related to ELI-002
Description: The safety of ELI-002 was monitored through adverse events, including those considered related to treatment by the investigator
Time Frame: Adverse events were collected through 28 days after the last dose
Population: All enrolled subjects were included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | ELI-002 2P Cohort 1 | ELI-002 2P Cohort 2 | ELI-002 2P Cohort 3 | ELI-002 2P Cohort 4 | ELI-002 2P Cohort 5
Number analyzed (Participants) | 3 | 6 | 5 | 5 | 6
Participants | 1 | 3 | 2 | 2 | 4

2. Secondary Outcome: The Proportion of Participants With Biomarker Reduction
Description: A biomarker reduction was any decrease from baseline in circulating tumor DNA (ctDNA) and/or serum tumor antigen levels (carbohydrate antigen 19-9 [CA19-9] or carcinoembryonic antigen [CEA]).
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | ELI-002 2P Cohort 1 | ELI-002 2P Cohort 2 | ELI-002 2P Cohort 3 | ELI-002 2P Cohort 4 | ELI-002 2P Cohort 5
Number analyzed (Participants) | 3 | 6 | 5 | 5 | 6
Participants | 2 | 5 | 4 | 4 | 6

3. Secondary Outcome: The Proportion of Participants With Biomarker Clearance
Description: Biomarker clearance was defined as no detectable ctDNA, CA19-9, or CEA at post-treatment time points.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | ELI-002 2P Cohort 1 | ELI-002 2P Cohort 2 | ELI-002 2P Cohort 3 | ELI-002 2P Cohort 4 | ELI-002 2P Cohort 5
Number analyzed (Participants) | 3 | 6 | 5 | 5 | 6
Participants | 1 | 2 | 1 | 1 | 1

4. Secondary Outcome: The Proportion of Participants With Biomarker Reduction by Biomarker Type
Description: A biomarker reduction was any decrease from baseline in ctDNA and/or serum tumor antigen levels (CA19-9 or CEA).
Time Frame: 6 months
Population: All enrolled subject by biomarker type at baseline
Measure: Count of Participants; unit: Participants
Groups:
- ctDNA Group: The ctDNA Group included subjects with detectable ctDNA at baseline.
- Serum Tumor Biomarker Group: The Serum Tumor Biomarker Group included subjects who did not have detectable ctDNA at baseline, but did have either detectable CA19-9 or CEA.
Arm/Group | ctDNA Group | Serum Tumor Biomarker Group
Number analyzed (Participants) | 13 | 12
Participants | 12 | 9

5. Secondary Outcome: The Proportion of Participants With Biomarker Clearance by Biomarker Type
Description: Biomarker clearance was defined as no detectable ctDNA, CA19-9, or CEA at post-treatment time points
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | ctDNA Group | Serum Tumor Biomarker Group
Number analyzed (Participants) | 13 | 12
Participants | 6 | 0

ADVERSE EVENTS:
Time Frame: For each participant, adverse events were collected through 28 days after the last dose. The last planned dose was at approximately 9 months.
Arm/Group | ELI-002 2P Cohort 1 | ELI-002 2P Cohort 2 | ELI-002 2P Cohort 3 | ELI-002 2P Cohort 4 | ELI-002 2P Cohort 5
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/6 | 0/5 | 0/5 | 0/6
Serious Adverse Events (participants affected / at risk) | 1/3 | 0/6 | 0/5 | 0/5 | 1/6
Other Adverse Events (participants affected / at risk) | 3/3 | 5/6 | 4/5 | 4/5 | 5/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ELI-002 2P Cohort 1 (N=3) | ELI-002 2P Cohort 2 (N=6) | ELI-002 2P Cohort 3 (N=5) | ELI-002 2P Cohort 4 (N=5) | ELI-002 2P Cohort 5 (N=6)
Abdominal wall haematoma (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ELI-002 2P Cohort 1 (N=3) | ELI-002 2P Cohort 2 (N=6) | ELI-002 2P Cohort 3 (N=5) | ELI-002 2P Cohort 4 (N=5) | ELI-002 2P Cohort 5 (N=6)
Anaemia (Blood and lymphatic system disorders) | 2 | 0 | 1 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Dermoid cyst (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 1
Hypermobility syndrome (Congenital, familial and genetic disorders) | 0 | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 2
Anal fissure (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Gastric ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Gingival pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0
Proctalgia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Catheter site pain (General disorders) | 0 | 1 | 0 | 0 | 0
Chills (General disorders) | 0 | 0 | 0 | 0 | 1
Fatigue (General disorders) | 1 | 2 | 2 | 1 | 1
Injection site erythema (General disorders) | 0 | 1 | 0 | 0 | 0
Injection site induration (General disorders) | 0 | 1 | 0 | 0 | 0
Injection site swelling (General disorders) | 0 | 1 | 0 | 0 | 0
Localised oedema (General disorders) | 0 | 0 | 0 | 0 | 1
Malaise (General disorders) | 1 | 1 | 0 | 0 | 1
Nodule (General disorders) | 0 | 0 | 0 | 0 | 1
Pneumonia cryptococcal (General disorders) | 0 | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 1 | 0 | 0 | 0
COVID-19 (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Herpes simplex reactivation (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Weight decreased (Investigations) | 0 | 1 | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Hyperglycaemai (Metabolism and nutrition disorders) | 0 | 0 | 2 | 2 | 2
Hyperphospataemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 1
Muscle spasm (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 2 | 1 | 0 | 0 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 1 | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 1 | 1 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 2
Pelvic pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 2 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Sensitive skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Hot flush (Vascular disorders) | 0 | 1 | 0 | 0 | 1
Peripheral arterial occlusive disease (Vascular disorders) | 0 | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2023-08-07): https://cdn.clinicaltrials.gov/large-docs/17/NCT04853017/Prot_000.pdf
  • Statistical Analysis Plan (2024-09-16): https://cdn.clinicaltrials.gov/large-docs/17/NCT04853017/SAP_001.pdf